CLINICAL TRIAL: NCT05586711
Title: Effects of Local Dehydroepiandrosterone (DHEA) and Estradiol on Moderate to Severe Dyspareunia, a Symptom of Vulvovaginal Atrophy in Postmenopausal Women - a Randomized, Controlled Study
Brief Title: Local DHEA and Estradiol on Dyspareunia in Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Angelica Lindén Hirschberg (Other)
Responsible Party: Sponsor-Investigator, Angelica Lindén Hirschberg, Professor, MD, PhD, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-003254-76
Record Dates: First submitted 2022-10-09; First posted 2022-10-19 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Vulvovaginal Atrophy; Genitourinary Syndrome of Menopause
Keywords: Vulvovaginal atrophy; Genitourinary Syndrome of Menopause

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal estradiol 10 μg (Active Comparator)
  Interventions: Drug: vaginal estradiol 10 μg
- Vaginal DHEA 6,5 mg (Active Comparator)
  Interventions: Drug: vaginal DHEA 6.5 mg

INTERVENTIONS:
Drug: vaginal estradiol 10 μg — Vagifem® (estradiol), vaginal tablets
  Arms: Vaginal estradiol 10 μg
Drug: vaginal DHEA 6.5 mg — Intrarosa® (dehydroepiandrosterone; DHEA; prasterone), pessaries
  Arms: Vaginal DHEA 6,5 mg

SUMMARY:
Vulvovaginal atrophy (VVA) is a condition characterized by vaginal dryness, itching, burning, irritation and dyspareunia. The condition is mainly due to estrogen deficiency and is common during and after menopause. Furthermore, androgens may have an important function in these symptoms. The purpose of the study is to compare vaginal estrogen with vaginal dehydroepiandrosterone (DHEA, an androgen precursor) on dyspareunia (primary outcome), a symptom of VVA in postmenopausal women. Secondary outcomes are total symptom score of VVA (vaginal dryness, irritation/itching, maturation index, pH), clinical signs of VVA, sexual function, urogenital symptoms, vaginal histomorphology, sex hormone levels and short-term safety. The hypothesis of the study is that the treatments will have a similar effect on dyspareunia while DHEA, through local androgenic effects (eg growth of muscle tissue and nerve density in the vaginal wall), may be more effective in treating other related symptoms such as sexual dysfunction. 170 postmenopausal women will be randomly assigned to treatment with either vaginal estrogen (Vagifem) or vaginal DHEA (Intrarosa). The women are examined at the start of the study, after 4 weeks of daily application and after another 8 weeks of treatment with twice a week application of the vaginal treatment. The study is expected to provide increased knowledge about the effect of the treatments of VVA in postmenopausal women as well as whether vaginal DHEA has additional positive effects on sexual function compared to vaginal estrogen.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (non-hysterectomized or hysterectomized) must satisfy either: a) No menses for at least one year for non-hysterectomized women, or b) Follicle stimulating hormone (FSH) levels >40 IU/L
* Women who have self-identified at screening and baseline (Day 1) as experiencing moderate to severe dyspareunia, using VASQ questionnaire (section 1)
* Between 40 and 80 years of age
* Body mass index (BMI) 19-35
* Women having a vaginal pH above 5 at screening and baseline (Day 1)
* Women who currently have intercourse or other sexual activity, at least once a month, with a partner
* Normal mammogram within 12 months (of Day 1)
* A normal PAP smear (which includes inflammatory changes) within the last 12 months (of Day 1) for both non-hysterectomized and hysterectomized women.
* Understands Swedish and is willing to participate in the study and sign an informed consent

Exclusion Criteria:

* Undiagnosed abnormal vaginal bleeding
* Previous diagnosis of cancer, except skin cancer (non-melanoma)
* Lichen Sclerosis and other pathological conditions in vulva and/or vagina
* Active or history of thromboembolic disease
* Clinically significant metabolic or endocrine disease (including diabetes mellitus) not controlled by medication
* Oral estrogen, progestin or DHEA exposure or intrauterine progestin therapy in the 8 weeks prior to baseline assessments (screening visit)
* Vaginal hormonal products (rings, creams, gels or tablets) or transdermal estrogen alone or estrogen/progestin products in the 4 weeks prior to baseline assessments (screening visit)
* Use of testosterone or other anabolic steroid within 6 months prior to screening visit
* Natural oral estrogenic products in the 4 weeks prior to baseline assessments
* Confirmed clinically significant depression (not controlled by standard therapy) or confirmed history of severe psychiatric disturbance
* The administration of any investigational drug within 30 days of screening visit

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Dyspareunia, a symptom of VVA in postmenopausal women | Primary endpoint will be evaluated as change in dyspareunia (VASQ section 1) from baseline to Week 12
  Patient reports in the Vaginal Atrophy Symptoms Questionnaire (VASQ, section 1). A 4-point scale, where a higher point means more symptoms.

SECONDARY OUTCOMES:
Total symptom score of VVA | Change from baseline to Week 4 and 12
  Vaginal dryness and irritation/itching (VASQ, section 2 and 3, a 4-point scale, where a higher point means more symptoms)
Clinical signs of VVA | Change from baseline to Week 4 and 12
  Examination of vaginal atrophy symptoms (VAX). A 4-point scale, where a higher point means more symptoms.
Sexual function | Change from baseline to Week 4 and 12
  Profile of Female Sexual Function (PFSF) and its seven domains desire, arousal, orgasm, pleasure, concern, responsiveness and self-image (range from 0 to 100, where a lower score means more dysfunction)
Urinary incontinence | Change from baseline to Week 4 and 12
  The Incontinence Impact Questionnaire (IIQ-7, a 4-point scale, where a higher point means more symptoms)
Histomorphology of the vaginal wall | Change from baseline to Week 4 and 12
  Histomorphology (thickness of epithelium, lamina propria and muscle layer in vaginal biopsies)
Sex hormone levels | Change from baseline to Week 4 and 12
  Sex hormone levels (estradiol and testosterone)

OTHER OUTCOMES:
Sexual activity | Change from baseline to Week 4 and 12
  Sexual activity log (SAL, the number of satisfying sexual episodes over a 1-week period)
Sexual distress | Change from baseline to Week 4 and 12
  the Personal Distress Scale (PDS, 0 [no distress] to 100 [maximum distress]).
Urogenital distress | Change from baseline to Week 4 and 12
  Urogenital Distress Inventory (UDI-6, a 4-point scale, where a higher point means more symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden